CLINICAL TRIAL: NCT01989806
Title: Investigation on the Effect of Robotic-assisted Body Weight Supported Treadmill Training on Walking and Cardiopulmonary Recovery in Patients Suffering From Incomplete Spinal Cord Injury
Brief Title: Robotic-assisted Locomotor Training on Mobility and Cardiopulmonary Function in Patients Suffering From Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kowloon Hospital, Hong Kong (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Mr. Cheung Yu Yeung, Physiotherapist II, Kowloon Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCI-1
Record Dates: First submitted 2013-11-08; First posted 2013-11-21 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Spinal Cord Injury
Keywords: Spinal cord injury; robotic; locomotion
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Robotic-assisted body weight supported treadmill training (Active Comparator): Robotic assisted body weight supported treadmill training with conventional PT training
  Interventions: Device: Robotic-assisted body weight supported treadmill training (Lokomat V6, Hocoma AG, Switzerland)
- Passive lower limbs mobilization training (Placebo Comparator): Passive lower limbs mobilization training with conventional PT training
  Interventions: Device: Passive lower limbs mobilization training (Motomed Vivo 2, RECK, Germany)

INTERVENTIONS:
Device: Robotic-assisted body weight supported treadmill training (Lokomat V6, Hocoma AG, Switzerland)
  Arms: Robotic-assisted body weight supported treadmill training
Device: Passive lower limbs mobilization training (Motomed Vivo 2, RECK, Germany)
  Arms: Passive lower limbs mobilization training

SUMMARY:
Evidences showed that patients suffering from spinal cord injury (SCI) have poor mobility and higher chance to develop cardiopulmonary diseases, which leads to poor quality of life and shorter life expectancy. Different modalities were developed aiming at mobility restoration in SCI patients and robotic assisted body weight supported treadmill training is one of the latest technique in recent years. Yet there are scarce studies to investigate its effectiveness. The purpose of this study is to investigate the effectiveness of robotic-assisted body weight supported treadmill training on mobility and cardiopulmonary function of patients suffering from SCI by a randomized controlled trial.

80 patients suffering from incomplete SCI will be recruited for an 8-week training program. They will be randomized into either robotic assisted body weight supported treadmill training group or passive lower limb mobilization training group. The training effects will be measured by Walking Index for Spinal Cord Injury version II, lower extremity motor score, lower limb Modified Ashworth Scale, robotic gait system, gait analysis and gas analysis under sub maximal exercise stress test.

Through the study, we intent to find the effectiveness of robotic-assisted body weight support treadmill training on walking and cardiopulmonary recovery with patients suffering from incomplete spinal cord injury.

The hypothesis of the study is:

Compared to the control group, robotic-assisted body weight supported treadmill training leads to a greater improvement in walking ability and cardiopulmonary functioning.

DETAILED DESCRIPTION:
Participants will be recruited from the spinal cord rehabilitation unit of Physiotherapy Department of Kowloon Hospital. Subjects will be allocated into intervention group or control group by using sealed envelope and they will be blinded for their group allocation. All participants will undergo standard physiotherapy program, including mobilization and strengthening exercise of limbs, trunk stabilization training, wheelchair maneuver training and overground walking training. Based on this standard training program twice per week, 60 minutes per session, participants will receive an additional 30 minutes (exclude set-up time) of robotic-assisted body weight supported treadmill training (BWSTT) or control training based on their group allocation 3 times for 8 week. EMG biofeedback system will be applied to bilateral vastus lateralis muscles during training with audio feedback to promote active participation.

Outcome measures will be collected before the intervention and the subjects will be reassessed after finishing their 8 weeks of intervention. Outcome measures include Walking Index for Spinal Cord Injury version II, Spinal Cord Independence Measure version III, lower extremity motor score, Modified Ashworth Scale, L-stiff and L-force measured by Lokomat system, VO2 maximum, spirometry, and gait analysis (walking speed, heel-heel base support,bilateral stance duration, bilateral symmetry) The result of this study will provide useful information to enhance the clinical effectiveness of the management for spinal cord injury with the use of robotic assisted body weight supported treadmill training.

ELIGIBILITY:
Inclusion Criteria:

* adult patient with age 18 or above
* suffering from incomplete spinal cord injury with classification B, C or D under the International Standards for Neurological Classification of Spinal Cord Injury (ISNSCI)
* lesion level above or at T12; acquired the injury not more than 24 months at the time of recruitment
* traumatic or non-traumatic, non-progressive lesion
* able to tolerate standing on tilt-table in 90 degrees for more than 30 minutes
* able to walk with or without orthosis but requires manual assistance in walking.

Exclusion Criteria:

* fracture of spine or lower limbs which is not yet stabilized
* severe osteoporosis or at high risk of pathological fracture
* symptomatic postural hypotension; cardiac disease which is not recommended for moderate intensity exercise
* severe muscle spasticity over lower limbs
* severe lower limbs fixed contractures
* leg length discrepancy for more than 2 centimeters
* body weight exceeding 135 kilograms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in Walking Index for Spinal Cord Injury version II from baseline to 8 weeks | Baseline, 8 weeks
  A validated mobility independence assessment tool for spinal cord injury (SCI) population (Burns, Delparte, Patrick, Marino, & Ditunno, 2011). Subjects will be asked to walk on a 10-meter straight line and score will be given based on the use of walking aids, orthoses, manual assistance and distance covered.

OTHER OUTCOMES:
Change in Spinal Cord Independence Measure version III from baseline to 8 weeks | Baseline, 8 weeks
  A validated assessment tool for SCI patients (Catz et al., 2007) to measure performance in different aspects, including self-care ability, respiratory and sphincter management and mobility.. For self-care and respiratory & sphincter domain, scoring will be given based on patient's subjective report while the mobility performance will be tested by the assessors.
Change in lower extremity motor score from baseline to 8 weeks | Baseline, 8 weeks
  The sum of muscle power of the 5 key muscles of lower limb. Manual muscle testing will be adopted in testing the muscle power and the grading will be based on the Medical Research Council scale for muscle strength.
Change in Modified Ashworth Scale from baseline to 8 weeks | Baseline, 8 weeks
  Hip and knee flexors and extensors will be tested. Subjects will be asked to relax during lying supine and assessor will passively move the limbs in fast speed. Scoring will be given based on the occurrence and quality of resistance.
Change in L-force from baseline to 8 weeks | Baseline, 8 weeks
  Strength will be assessed by L-force function which is installed in Lokomat system. subjects will be asked to perform isometric muscle contraction of hips and knees, the sensors in orthoses will measure the force exerted on it and record the result.
Change in walking quality from baseline to 8 weeks | Baseline, 8 weeks
  Walking speed, heel-heel base of support, bilateral legs stance duration and bilateral symmetry will be assessed by gait analysis system (GAITRite System, CIR Systems, Inc., US) . Subjects will be asked to walk on a pressure-detectable walkway, which is connected to a computer system. Assistance as well as orthoses will be provided based on subject's own choice. Two meters of acceleration distance will be provided before the subject walk onto the walkway while another two meters of deceleration distance will be provided so as to ensure that subjects walk with their fastest comfortable speed on the whole track of walkway. Bilateral symmetry will be assessed by the stride length ratio as well as stance phase duration ratio of the weak limb to strong limb, where the strong limb is defined as the one with higher score in lower extremity motor score.
Change in maximal oxygen consumption from baseline to 8 weeks | Baseline, 8 weeks
  For cardiopulmonary functioning, the subject will be asked to perform upper limb ergometry (Endorphin's 300 e2 resistance system, Endorphin Corporation, US) with a gas analysis system (Fitmate pro, COSMED, Italy). Subjects will wear a mask connecting to the gas analysis system and they will be asked to perform the upper limb ergometry with the following protocol: 1 minute of rest following with 1 minute of warm-up using the least resistance, then the resistance will be increased by 1 level per 1 minute time. The test will be stopped when the heart rate reaches 85% of maximal heart rate, or the subject cannot further tolerate the test. Maximal oxygen consumption will be recorded for further analysis.
Change in L-stiff from baseline to 8 weeks | Baseline, 8 weeks
  Stiffness will be assessed by L-stiff function, which subjects will be asked to keep relaxing on the system while the Lokomat system performs passive limbs movement at different speed. The torque during movement will be detected by the sensors in the orthoses and recorded the result.
Spirometry | Baseline, 8 weeks
  Spirometry will be used to assess the respiratory function of subjects. Subjects will be asked to perform a forced and prolonged expiration via mouth piece which connecting to a spirometer (Pony FX, COSMED, Italy) followed with a forced inspiration. A soft clip will be applied to subject's nose to minimize air leak from nose during test. Peak expiratory flow (PEF), forced expiratory flow rate in first second (FEV1) and forced vital capacity (FVC) will be assessed. 3 trials will be performed with 1 minute rest interval to prevent hyperventilation and the average value of the 3 trials will be recorded for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Cheung Yu Yeung E, BSc, Principal Investigator — Kowloon Hospital, Hong Kong
Locations (1):
- Physiotherapy Department, Kowloon Hospital, Hong Kong, China

REFERENCES:
- [Derived] Cheung EYY, Yu KKK, Kwan RLC, Ng CKM, Chau RMW, Cheing GLY. Effect of EMG-biofeedback robotic-assisted body weight supported treadmill training on walking ability and cardiopulmonary function on people with subacute spinal cord injuries - a randomized controlled trial. BMC Neurol. 2019 Jun 24;19(1):140. doi: 10.1186/s12883-019-1361-z. PMID 31234791